CLINICAL TRIAL: NCT04007900
Title: Positive Affect Treatment (PAT) to Target Reward Mechanisms in Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSYCH-2018-27082
Record Dates: First submitted 2019-06-07; First posted 2019-07-05 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Anorexia Nervosa; Anorexia
Keywords: positive affect treatment
MeSH Terms: conditions — Anorexia Nervosa; Anorexia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Affect Treatment (Experimental): Individuals randomized to the intervention will participate in 20 therapy visits. Before each therapy visit, the participant will meet briefly with a member of the research staff, who will measure weight (blind to the participant) and administer the CHEDS, PANAS, and a pre-session feedback form that will assess how helpful the skills learned in the prior session had been over the past week. After the session, the participant will complete the post-session feedback form, which will assess how helpful the skills he or she perceived the skills from this session to be. These procedures will take approximately 10 minutes. Each intervention session will take approximately 50 minutes to complete. Therefore, each intervention visit will be approximately 1 hour long. Therapy sessions will take place either in the private office of a study therapist or in a consultation room of the Ambulatory Research Center.
  Interventions: Behavioral: Positive Affect Treatment
- Waitlist (No Intervention): For participants randomized to the waitlist control, the opportunity will be offered to participate in the intervention following the second assessment (20 weeks following their Baseline assessment).

INTERVENTIONS:
Behavioral: Positive Affect Treatment — PAT was designed as a 15-week intervention delivered in 3 modules. Module 1 (Pleasant Events Scheduling) uses behavioral activation methods to enhance positive experiencing before, during, and after rewarding events. Module 2 (Attending to the Positive) applies cognitive training techniques to promote shifting attention towards rewarding aspects of daily situations and to learn behavior mood associations. Module 3 (Cultivating the Positive) uses mindfulness approaches to foster reward experiencing. Treatment length has been expanded to 20 sessions to enhance the suitability of the intervention for AN and target the reward mechanisms that characterize AN. Additional adaptations include: 1) An emphasis on a mindful balance between reward and inhibition; 2) Additional module on shifting attention away from AN-specific rewards; 3) Addition of exercises to work towards long-term life goals and enhance healthy experiences; and 4) Further focus on navigating social rewards.
  Arms: Positive Affect Treatment

SUMMARY:
The goal of the proposed research is to determine the extent to which Positive Affect Treatment (PAT), a novel treatment targeting reward mechanisms, can effectively target the psychological reward deficits that maintain anorexia nervosa (AN), and thus improve clinical symptoms.

DETAILED DESCRIPTION:
Anorexia Nervosa is a serious disorder associated with high medical and psychiatric morbidity, poor quality of life, and the highest mortality rate of any psychiatric illness. Although many individuals with AN ultimately achieve remission, this process of recovery is slow, with only about 1/3 of individuals recovering in the first decade of illness, and is not always associated with an enhanced quality of life. Further, a substantial portion of those with AN do not recover; 20-30% of affected individuals maintain a chronic illness course or die prematurely. Interventions that enhance the probability of long-term remission from adult AN are lacking. Efficacious outpatient treatments have not been identified and, although inpatient treatment can restore healthy weight, up to 50% of patients with AN relapse within a year of discharge. This paucity of effective treatment may be due to existing interventions not targeting key mechanisms of the disorder. Advances in neuroscience have contributed promising insights about the processes that promote AN symptoms. However, these findings have not been adequately integrated into treatment for AN. It is critical that future treatment development utilize emerging research on the mechanisms of AN to develop more effectively targeted interventions. The goal of the proposed research is to determine the extent to which Positive Affect Treatment (PAT), a novel treatment targeting reward mechanisms, can effectively target the psychological reward deficits that maintain anorexia nervosa (AN), and thus improve clinical symptoms. To this end, we propose a small, randomized, wait-list controlled pilot trial of PAT adapted for AN (PAT-AN) to achieve the following aims: To asses the feasibility and acceptability of PAT-AN among individuals with AN and to obtain initial data regarding the potential efficacy of PAT-AN compared to waitlist control on measures of clinical outcome and putative reward mechanisms in AN to inform a future larger randomized, controlled trial of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of AN (established by the adapted MINI)
* Ability to read and speak in English
* Involvement in ongoing oversight with a primary physical or mental health provider as defined by:

  1. Identification by the participant of a physical or mental health provider (e.g., physician, psychiatrist, psychologist, masters level social worker, licensed professional clinical counselor, licensed marriage and family therapist) who will serve as the primary provider throughout the study
  2. Willingness to sign a Release of Information that gives the study therapist the right to discuss any change in medical or psychiatric stability or other health concerns with the participant's identified primary provider.

Exclusion Criteria:

* Medical instability according to standard guidelines and medical staff judgment
* Acute suicidality, current substance use disorder, psychosis, or mania requiring specialized treatment
* Lacking capacity to consent
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Efficacy: Change in BMI | 20-weeks
  Body mass index (BMI) will be calculated based on height and weight measure by a stadiometer and calibrated scale during a medical examination. Change in BMI (kg/m2) will be calculated from baseline to 20-weeks. Increase in BMI in the treatment group vs control will be considered a measure of efficacy of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States